CLINICAL TRIAL: NCT06326931
Title: A Prospective, Randomized Comparison of Thermal Pulsation Versus Warm Compress Treatment for Signs and Symptoms of Meibomian Gland Dysfunction
Brief Title: Thermal Pulsation Versus Warm Compress Treatment for Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jacksoneye (Other)
Responsible Party: Principal Investigator, Melissa Bollinger, OD, FAAO, Principle Investigator, Jacksoneye
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JE001
Record Dates: First submitted 2024-03-18; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: The clinician evaluating MGS score was masked to subject treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Thermal pulsation group (Experimental): Group treated in both eyes with a single Systane iLux thermal pulsation treatment
  Interventions: Device: thermal pulsation
- Warm compress group (Active Comparator): Group treated in both eyes with 10 minute application of Bruder warm compress mask, twice daily for 8 weeks
  Interventions: Other: warm compress

INTERVENTIONS:
Device: thermal pulsation — Single, in-office bilateral treatment with Systane iLux thermal pulsation
  Other Names: Systane iLux
  Arms: Thermal pulsation group
Other: warm compress — Twice daily, 10-minute at-home treatment with Bruder warm compress mask for 8 weeks
  Other Names: Bruder mask
  Arms: Warm compress group

SUMMARY:
This study aimed to assess the treatment outcome differences between a single, in-office bilateral treatment with the thermal pulsation system and twice-daily, 10-minute applications of the warm compress mask at home for 8 weeks.

DETAILED DESCRIPTION:
This prospective, single-center, single-masked, randomized, controlled clinical trial compared the Systane iLux handheld thermal pulsation system with a warm compress mask (Bruder Moist Heat Eye Compress, Bruder Healthcare, Alpharetta, GA, USA) for the treatment of meibomian gland dysfunction (MGD).

Subjects aged 18 or older were randomized 1:1 to either a single in-office thermal pulsation treatment or twice-daily use of the warm compress mask, with both eyes undergoing the same treatment. Enrollment criteria included Ocular Surface Disease Index (OSDI) score >23, total meibomian gland secretion (MGS) score < or =12 in the lower lid of each eye, and tear break-up time (TBUT) < 10 seconds. TBUT, MGS, and corneal staining scores were evaluated at baseline, 2 weeks, and 8 weeks. Symptoms were evaluated using the OSDI questionnaire at baseline, 2 weeks, and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* history of self-reported dry eye symptoms for 3 months prior to study enrollment
* baseline OSDI score of 23 or greater (
* MGS score of 12 ior less in the lower eyelid of each eye
* TBUT <10 seconds
* willing and able to abstain from using any new ocular lubricants

Exclusion Criteria:

* diagnosis of thyroid dysfunction or rheumatoid arthritis
* history of laser-assisted in situ keratomileusis (LASIK); any other ocular surgery within the previous 12 months
* abnormal lid anatomy or active lid lesions
* use of topical glaucoma medications, medications affecting the central nervous system, or hormonal drugs within the previous month
* active ocular infection
* pterygium
* planned use of contact lenses, topical antibiotics, steroids, or immunomodulating drops
* CDVA worse than 0.2 logMAR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Change in MGS score for the worse eye | baseline to Week 8
  Change in MGS score for the worse eye

SECONDARY OUTCOMES:
Change in MGS score for the worse eye | baseline to Week 2
  Change in MGS score for the worse eye
Change in OSDI score | Baseline to Week 2
  Change in OSDI score
Change in OSDI score | Baseline to Week 8
  Change in OSDI score
Incidence of adverse events | 8 weeks
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bollinger, OD, FAAO, Principal Investigator — Jacksoneye
Locations (1):
- Jacksoneye, Lake Villa, Illinois, United States

IPD SHARING:
Plan to Share IPD: No